CLINICAL TRIAL: NCT02479204
Title: Single-center, Open-label, Randomized, Multiple-dose, Parallel-group Study to Investigate Safety and Effects on Heart Rate, Blood Pressure, and Pharmacokinetic Interactions of ACT-334441 Combined With Calcium-channel Blocker (Diltiazem) or Beta-blocker (Atenolol) Treatment in Healthy Subjects
Brief Title: Clinical Study to Investigate Safety and Effects on Heart Rate, Blood Pressure, and Pharmacokinetic Interactions of ACT-334441
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on results from the pilot phase, the study is terminated. No safety events leading to discontinuation were reported
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AC-064-102
Record Dates: First submitted 2015-06-17; First posted 2015-06-24 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2018-07

CONDITIONS: Healthy Subjects
Keywords: safety; heart rate; pharmacokinetics
MeSH Terms: interventions — Atenolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A ACT-334441 + atenolol (Experimental): 4 subjects will receive 50 mg of atenolol once daily for 6 days, and a concomitant single administration of ACT-334441 2 mg on Day 6
  Interventions: Drug: ACT-334441 2 mg; Drug: Atenolol
- Part A ACT-334441 + diltiazem (Experimental): 4 subjects will receive 240 mg of diltiazem once daily for 6 days, and a concomitant single administration of ACT-334441 2 mg on Day 6
  Interventions: Drug: ACT-334441 2 mg; Drug: Diltiazem ER
- Part B ACT-334441 + atenolol (Experimental): 12 subjects will receive 50 mg of atenolol (once daily) from day 1 to day 15, placebo once on day 6, and ACT-334441 4 mg (once daily) from day 8 to day 15
  Interventions: Drug: ACT-334441 4 mg; Drug: Placebo; Drug: Atenolol
- Part B ACT-334441 + diltiazem (Experimental): 12 subjects will receive 240 mg of diltiazem (once daily) from day 1 to day 15, placebo once on day 6, and ACT-334441 4 mg (once daily) from day 8 to day 15
  Interventions: Drug: ACT-334441 4 mg; Drug: Placebo; Drug: Diltiazem ER

INTERVENTIONS:
Drug: ACT-334441 2 mg — capsule containing ACT-334441 at a strength of 2 mg
  Arms: Part A ACT-334441 + atenolol; Part A ACT-334441 + diltiazem
Drug: ACT-334441 4 mg — capsule containing ACT-334441 at a strength of 4 mg
  Arms: Part B ACT-334441 + atenolol; Part B ACT-334441 + diltiazem
Drug: Placebo — ACT-33441-matching placebo
  Arms: Part B ACT-334441 + atenolol; Part B ACT-334441 + diltiazem
Drug: Atenolol — film-coated tablet containing atenolol at a strength of 50 mg
  Other Names: Tenormine
  Arms: Part A ACT-334441 + atenolol; Part B ACT-334441 + atenolol
Drug: Diltiazem ER — film-coated tablet containing diltiazem at a strength of of 120 mg
  Other Names: Bi-tildiem
  Arms: Part A ACT-334441 + diltiazem; Part B ACT-334441 + diltiazem

SUMMARY:
The aim of the study is to investigate the safety of the concomitant administration of ACT-334441 with cardiovascular drugs.

DETAILED DESCRIPTION:
The study will consist of two parts: a pilot part (Part A) that will be completed prior to the start of the main part (Part B). The Subjects who will participate in Part A are excluded from Part B.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Body mass index (BMI) between 18.0 and 30.0 kg/m2 (inclusive) at screening.
* Women of childbearing potential must have a negative pregnancy test and they must use reliable methods of contraception
* Healthy on the basis of physical examination,cardiovascular assessments and laboratory tests

Exclusion Criteria:

* Pregnant or lactating women
* Any contraindication to the study drugs
* History or presence of any disease or condition or treatment, which may put the subject at risk of participation in the study or may interfere with the absorption, distribution, metabolism or excretion of the study drugs
* Any clinically significant abnormalities in laboratory tests, vital signs, ECG variables and pulmonary variables
* Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-05-01 (Actual)

PRIMARY OUTCOMES:
PR intervals measured by 12-lead ECG (Part A + Part B) | Days 1 and 6 (Part A); Days 1, 6, 8, 9, 15, and 16 (Part B)
  Absolute PR intervals and corresponding changes from baseline at the different days of measurement
Heart rate (HR) measured by 12-lead ECG (PArt A + Part B) | Days 1 and 6 (Part A); Days 1, 6, 8, 9, 15, and 16 (Part B)
  Absolute heart rates at the different days of measurement
Hourly mean heart rate (HR) measured by 24-hour Holter ECG | Days 1 and 6 (Part A); Days 1, 6, 8, 9, 15, and 16 (Part B
  Absolute and change from baseline in hourly mean HR on each day of measurement

SECONDARY OUTCOMES:
Areas under the plasma concentration-time curves (AUC) for ACT-334441, diltiazem and atenolol (Part B) | Blood samples from Day 1 to Day 20 for the PK profile of diltiazem and atenolol, and from Day 8 to Day 21 for the PK profile of ACT-334441.
  AUCs will be calculated will be calculated according to the linear trapezoidal rule for the following periods: from zero to time t of the last measured concentration above the limit of quantification, from zero to 24h after study drug administration, from zero to infinity)
Maximum plasma concentration (Cmax) for ACT-334441, diltiazem and atenolol (Part B) | From Day 1 to Day 20 for diltiazem and atenolol; from Day 8 to Day 21 for ACT-33444.
  The measured individual concentrations of ACT-334441, diltiazem and atenolol will be used to obtain their respective Cmax
Time to reach the maximum plasma concentration (tmax) for ACT-334441, diltiazem and atenolol (Part B) | From Day 1 to Day 20 for diltiazem and atenolol; from Day 8 to Day 21 for ACT-33444
  The measured individual concentrations of ACT-334441, diltiazem and atenolol will be used to obtain their respective tmax
Terminal half-life [t(1/2)] of ACT-334441, diltiazem and atenolol (Part B) | From Day 1 to Day 20 for diltiazem and atenolol; from Day 8 to Day 21 for ACT-33444
  Time required for the plasma concentration of a drug to decrease by 50% in the final stage of its elimination
Trough plasma levels (Ctrough) of of ACT-334441, diltiazem and atenolol (Part B) | From Day 1 to Day 15 for diltiazem and atenolol; from Day 8 to Day 15 for ACT-33444
  Ctrough will be used to determine the attainment of steady state conditions
Number of subjects with adverse events as a measure of safety | From baseline to end of study [Day 20-23 (Part A), Day 556-59 (Part B)]
  An AE is defined as any unfavorable and unintended sign, including an abnormal laboratory finding, symptom or disease, that occurs during the course of the study, whether or not considered related to the study drug

OTHER OUTCOMES:
Lymphocyte count as a measure of immunomodulation (Part A + Part B) | Day 1, Day 6, Day 12 and Day 20 (Part A); Day 1 and Day 8 toDay 16 (Part B)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (1):
- BIOTRIAL, Rennes, France